CLINICAL TRIAL: NCT06132126
Title: A Single and Multiple-Ascending Dose Phase 1 Study to Assess the Safety, Tolerability, and Pharmacokinetics of LY3938577 in Healthy Participants and Participants With Type 2 Diabetes Mellitus
Brief Title: A Study to Investigate the Safety and Tolerability of LY3938577 in Healthy Participants and Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 18779; J4P-MC-IYAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Healthy; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LY3938577 (Part A) (Experimental): LY3938577 administered Subcutaneously (SC).
  Interventions: Drug: LY3938577
- Placebo (Part A) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo
- Insulin degludec (Part A) (Active Comparator): Insulin degludec administered SC.
  Interventions: Drug: Insulin degludec
- LY3938577 (Part B) (Experimental): LY3938577 administered SC.
  Interventions: Drug: LY3938577
- Insulin degludec (Part B) (Active Comparator): Insulin degludec administered SC.
  Interventions: Drug: Insulin degludec

INTERVENTIONS:
Drug: LY3938577 — Administered SC.
  Arms: LY3938577 (Part A); LY3938577 (Part B)
Drug: Placebo — Administered SC.
  Arms: Placebo (Part A)
Drug: Insulin degludec — Administered SC.
  Arms: Insulin degludec (Part A); Insulin degludec (Part B)

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of a single dose of LY3938577 in healthy participants and participants with Type 2 Diabetes Mellitus (T2DM) (Part A) and multiple doses of LY3938577 in participants with T2DM (Part B). The study will last approximately 6 weeks for Part A and approximately 10 weeks for Part B respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are overtly healthy as determined by medical evaluation (Part A)
* Participants with T2DM diagnosed greater than 1 year before enrollment (Part A and Part B)
* Have a body mass index within the range of 18.5 to less than or equal to (<=) 32 kilograms per square meter (kg/m²) for healthy participants and 18.5 to 40 kg/m² for T2DM participants.
* Male or female participants of nonchildbearing potential

Exclusion Criteria:

* Have proliferative retinopathy or maculopathy and/or severe neuropathy
* Have been treated with sulfonylurea, thiazolidinedione, alpha-glucosidase inhibitor, glucagon-like peptide-1 receptor agonist or Insulin within the previous 3 months
* Have received chronic systemic glucocorticoid therapy in the past 3 months
* Are currently enrolled in another clinical study trial involving medical research, or have participated within the last 30 days in a clinical study involving an investigational product.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Part A: Number of participants with one or more Adverse Event (s) (AEs), and Serious Adverse Event(s) (SAEs) considered by the investigator to be related to study drug administration | Baseline up to 16 days
  A summary of AEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module.
Part B: Number of participants with one or more Adverse Event (s) (AEs), and Serious Adverse Event(s) (SAEs) considered by the investigator to be related to study drug administration | Baseline up to 44 days
  A summary of AEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module.
Part A: Incidence of Hypoglycemia | Baseline up to 16 days
Part B: Incidence of Hypoglycemia | Baseline up to 44 days
Part A: Number of Participants With Clinically Significant Changes in Vital Signs | Baseline up to 16 days
Part B: Number of Participants With Clinically Significant Changes in Vital Signs | Baseline up to 44 days
Part A: Number of Participants With Clinically Significant Changes in Safety Laboratory Parameters | Baseline up to 16 days
Part B: Number of Participants With Clinically Significant Changes in Safety Laboratory Parameters | Baseline up to 44 days

SECONDARY OUTCOMES:
Part A and Part B: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) | Part A: Predose up to 16 Days and Part B: Predose up to 44 Days

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - CenExel ACT, Anaheim, California
  - Qps-Mra, Llc, Miami, Florida
  - Labcorp CRU, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Investigate the Safety and Tolerability of LY3938577 in Healthy Participants and Participants With Type 2 Diabetes Mellitus — https://trials.lilly.com/en-US/trial/436457.